CLINICAL TRIAL: NCT02371356
Title: Comparing Effectiveness of Treating Depression With & Without Comorbidity to Improve Fetal Health
Acronym: PCORIPTD
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CN-13-1650-H
Record Dates: First submitted 2015-01-28; First posted 2015-02-25 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Depression; Preterm Delivery
MeSH Terms: conditions — Depression; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Depressed, Medication only: Screen positive for depression and use only antidepressants during pregnancy
- Depressed, Psychotherapy only: Screen positive for depression and receive psychotherapy only.
- Depressed, Medication & Psychotherapy: Screen positive for depression and receive both antidepressants and psychotherapy.
- Depressed, untreated: Screen positive for depression and receive no treatment.
- Not depressed: Screen negative for depression and receive no treatment.

SUMMARY:
Depression during pregnancy is prevalent (15-20%) and has an adverse impact on fetal outcomes including preterm delivery (PTD) and low birthweight (LBW). Currently, significant confusion exists about if and how depression during pregnancy should be treated, given the unknown risk-benefit profiles of various treatments. We propose to conduct a two-stage prospective cohort study to determine if treating depression in pregnancy is effective in improving fetal outcomes, and which treatment is most effective: pharmacotherapy, psychotherapy or a combination. The risk-benefit of the treatments will be examined separately for two depression types: pregnant women with depression only and those with other psychiatric comorbidities to evaluate possible differences in treatment effectiveness between the two groups. Findings will provide answers to long standing stakeholder questions of how to treat depression in pregnancy and which treatment is most effective with the best risk-benefit profile in improving fetal outcomes. Selecting an effective treatment could reduce PTD or LBW, thus, reducing infant mortality and morbidity, and medical costs.

DETAILED DESCRIPTION:
Depression during pregnancy is prevalent (15-20%) and has an adverse impact on fetal outcomes including preterm delivery (PTD) and low birthweight (LBW). Currently, significant confusion exists about if and how depression during pregnancy should be treated, given the unknown risk-benefit profiles of various treatments. Kaiser Permanente Northern California has implemented a large scale universal peripartum depression screening program, annually screening more than 35,000 pregnant women. Taking advantage of this unique infrastructure, we propose to conduct a two-stage prospective cohort study to determine if treating depression in pregnancy is effective in improving fetal outcomes, and which treatment is most effective: pharmacotherapy, psychotherapy or a combination. The risk-benefit of the treatments will be examined separately for two depression types: pregnant women with depression only and those with other psychiatric comorbidities to evaluate possible differences in treatment effectiveness between the two groups. Stakeholders (patients, advocacy groups, and providers) are an integral part of the research team. Four cohorts with different treatment options including untreated will be formed within each depression type (with or without comorbidity): (A) "Antidepressant only": screen positive for depression and use only antidepressants during pregnancy; (B) "Psychotherapy only": screen positive and receive psychotherapy only; (C) "Combination therapy": screen positive and receive both antidepressants and psychotherapy; (D)"Untreated depression": screen positive and receive no treatment. A total of eight cohorts will be formed. A final cohort (E) "No depression": screen negative and receive no treatment, will be examined for baseline comparison. Information on depression treatment and PTD and LBW will be available for all participating women who will be followed until the end of pregnancy. Within each depression category, comparison of Cohort A, B & C to D, respectively, will determine if treating depression is effective. Pair-wise comparisons among Cohorts A, B & C will determine the comparative effectiveness of treatment regimens. Comparison of Cohort D to E provides baseline fetal risks of untreated depression. Findings will provide answers to long standing stakeholder questions of how to treat depression in pregnancy and which treatment is most effective with the best risk-benefit profile in improving fetal outcomes. Selecting an effective treatment could reduce PTD or LBW, thus, reducing infant mortality and morbidity, and medical costs.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser member
* Pregnant

Exclusion Criteria:

* Not a member of Kaiser Permanente
* Not pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant KPNC members who have been screened as part of KPNC's peripartum depression screening program, assigned to cohorts according to depression and treatment status.
Sampling Method: Non-Probability Sample
Enrollment: 91084 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01-31 (Actual); Study Completion 2019-04-30 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Depressed: Screen negative for depression and received no treatment
Period: Overall Study
Arm/Group | Depressed, Medication Only | Depressed, Psychotherapy Only | Depressed, Medication & Psychotherapy | Depressed, Untreated | Not Depressed
Started | 1320 | 7354 | 2804 | 7423 | 72183
Completed | 1320 | 7354 | 2804 | 7423 | 72183
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depressed, Medication Only | Depressed, Psychotherapy Only | Depressed, Medication & Psychotherapy | Depressed, Untreated | Not Depressed | Total
Number analyzed (Participants) | 1320 | 7354 | 2804 | 7423 | 72183 | 91084
Age, Customized [Count of Participants; unit: Participants]
  Maternal Age: 18-24 years | 156 | 1792 | 400 | 1123 | 8987 | 12458
  Maternal Age: 25-34 years | 721 | 4117 | 1654 | 4440 | 46148 | 57080
  Maternal Age: 35+ years | 443 | 1445 | 750 | 1860 | 17048 | 21546
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1320 | 7354 | 2804 | 7423 | 72183 | 91084
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Maternal Race/ethnicity: White | 813 | 2638 | 1610 | 2257 | 26385 | 33703
  Maternal Race/ethnicity: Asian | 103 | 1147 | 165 | 1957 | 19697 | 23069
  Maternal Race/ethnicity: African-American | 55 | 945 | 248 | 577 | 3773 | 5598
  Maternal Race/ethnicity: Hispanic | 283 | 2200 | 621 | 2208 | 18545 | 23857
  Maternal Race/ethnicity: Other/multiple/unknown | 66 | 424 | 160 | 424 | 3783 | 4857
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1320 | 7354 | 2804 | 7423 | 72183 | 91084

OUTCOME MEASURES:

1. Primary Outcome: Preterm Delivery
Description: Delivery prior to 37 completed weeks of gestational age
Time Frame: Through the end of pregnancy, an average of 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Depressed, Medication Only | Depressed, Psychotherapy Only | Depressed, Medication & Psychotherapy | Depressed, Untreated | Not Depressed
Number analyzed (Participants) | 1320 | 7354 | 2804 | 7423 | 72183
Participants
  Preterm | 139 | 556 | 272 | 569 | 4164
  Not preterm | 1181 | 6798 | 2532 | 6854 | 68019

2. Primary Outcome: Low Birth Weight
Description: Birth weight <2500 grams
Time Frame: Through the end of pregnancy, an average of 40 weeks
Population: Those with missing birth weight information were excluded from the analysis of low birth weight
Measure: Count of Participants; unit: Participants
Arm/Group | Depressed, Medication Only | Depressed, Psychotherapy Only | Depressed, Medication & Psychotherapy | Depressed, Untreated | Not Depressed
Number analyzed (Participants) | 1308 | 7251 | 2778 | 7310 | 72073
Participants
  Low birth weight | 82 | 408 | 158 | 385 | 3154
  Not low birth weight | 1226 | 6843 | 2620 | 6925 | 68919

ADVERSE EVENTS:
Time Frame: Overall Study: Through the end of pregnancy, an average of 40 weeks
Arm/Group | Depressed, Medication Only | Depressed, Psychotherapy Only | Depressed, Medication & Psychotherapy | Depressed, Untreated | Not Depressed
All-Cause Mortality (participants affected / at risk) | 0/1320 | 0/7354 | 0/2804 | 0/7423 | 0/72183
Serious Adverse Events (participants affected / at risk) | 0/1320 | 0/7354 | 0/2804 | 0/7423 | 0/72183
Other Adverse Events (participants affected / at risk) | 0/1320 | 0/7354 | 0/2804 | 0/7423 | 0/72183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02371356/Prot_SAP_000.pdf